CLINICAL TRIAL: NCT00003050
Title: Weekly Paclitaxel During Radiation Therapy for Locally Advanced Breat Cancer
Brief Title: Radiation Therapy Plus Paclitaxel in Treating Patients With Stage IIB or Stage III Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000065692 (1B-97-2); LAC-USC-1B972; NCI-G97-1304
Record Dates: First submitted 1999-11-01; First posted 2004-07-30 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; Doxorubicin; Paclitaxel; Tamoxifen; Surgical Procedures, Operative; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: paclitaxel
Drug: tamoxifen citrate
Procedure: surgical procedure
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with radiation therapy may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of radiation therapy plus paclitaxel in treating patients with stage IIB or stage III breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the safety and feasibility of twice a week paclitaxel and radiation therapy in patients with locally advanced breast cancer. II. Determine the pathological effects of paclitaxel and radiation in locally advanced breast cancer.

OUTLINE: This is a nonrandomized, dual institution study. Patients receive paclitaxel IV over 1 hour twice a week for a total of 8 weeks. This is started within 1 week of a tumor biopsy. Patients receive radiotherapy 5 days/week for 5.0 weeks within 1 week of the first paclitaxel dose. Operable patients who have progressive disease with the above therapy undergo a modified radical mastectomy (MRM), then receive 4 courses of doxorubicin IV and cyclophosphamide IV, administered once every 21 days. Inoperable patients receive this same chemotherapy regimen, then are reevaluated for surgery. Patients who have stable disease or who respond to the paclitaxel/radiation regimen undergo a MRM, then receive 4 courses of doxorubicin IV and paclitaxel IV (over 3 hours) once every 21 days. All patients with hormone receptor positive tumors receive tamoxifen for 5 years after all other therapy is completed.

PROJECTED ACCRUAL: A total of 40 patients (20 patients per institution) will be accrued over 18- 24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven, untreated, locally advanced breast cancer; stage IIB (T3 N0), IIIA, or IIIB Measurable disease Not inflammatory breast cancer or other stage IIB (T2 N1) No distant metastases except for positive ipsilateral supraclavicular nodes

PATIENT CHARACTERISTICS: Age: Over 18 Performance status: ECOG 0-1 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: Not pregnant Fertile patients must use effective contraception during and 6 months after treatment Medically and psychologically stable

PRIOR CONCURRENT THERAPY: No prior therapy of any type

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 1997-04; Primary Completion 2000-03 (Actual); Study Completion 2000-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darcy V. Spicer, MD, Study Chair — University of Southern California
Locations (2):
- United States (2):
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Mayo Clinic Jacksonville, Jacksonville, Florida

REFERENCES:
- [Result] Adams S, Chakravarthy AB, Donach M, Spicer D, Lymberis S, Singh B, Bauer JA, Hochman T, Goldberg JD, Muggia F, Schneider RJ, Pietenpol JA, Formenti SC. Preoperative concurrent paclitaxel-radiation in locally advanced breast cancer: pathologic response correlates with five-year overall survival. Breast Cancer Res Treat. 2010 Dec;124(3):723-32. doi: 10.1007/s10549-010-1181-8. Epub 2010 Sep 29. PMID 20878462
- [Result] Formenti SC, Volm M, Skinner KA, Spicer D, Cohen D, Perez E, Bettini AC, Groshen S, Gee C, Florentine B, Press M, Danenberg P, Muggia F. Preoperative twice-weekly paclitaxel with concurrent radiation therapy followed by surgery and postoperative doxorubicin-based chemotherapy in locally advanced breast cancer: a phase I/II trial. J Clin Oncol. 2003 Mar 1;21(5):864-70. doi: 10.1200/JCO.2003.06.132. PMID 12610186
- [Result] Formenti SC, Symmans WF, Volm M, Skinner K, Cohen D, Spicer D, Danenberg PV. Concurrent paclitaxel and radiation therapy for breast cancer. Semin Radiat Oncol. 1999 Apr;9(2 Suppl 1):34-42. PMID 10210538